CLINICAL TRIAL: NCT04132011
Title: Examining the Relationship Amongst Opioid Subjective Effects and Pharmacokinetics of Extended Release Opioids at Shortened Dosing Intervals in Patients With Chronic Pain: a Randomized, Blinded, N-of-1 Case Series Feasibility Study
Brief Title: Dosing Intervals of Opioid Medication for Chronic Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No recruitment (Feasibility study).
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Society of Hospital Pharmacists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-6180
Record Dates: First submitted 2019-10-02; First posted 2019-10-18 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2019-09

CONDITIONS: Chronic Pain
Keywords: opioid
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Feasibility study of an n-of-1, within-subject, crossover, randomized, double blind, placebo controlled case series
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shortened interval extended release opioid (Active Comparator): Extended release opioid, individualized total daily dose, dosing intervals less than every 12 hours.
  Interventions: Drug: Extended Release Opioid Formulation, Shortened Intervals; Drug: Placebo oral tablet
- Standard interval extended release opioid (Active Comparator): Extended release opioid, individualized total daily dose, dosing intervals every 12 hours
  Interventions: Drug: Extended Release Opioid Formulation, Standard intervals; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Extended Release Opioid Formulation, Shortened Intervals — Extended release opioid, individualized total daily dose, dosing interval is less than every 12 hours
  Other Names: Hydromorphone extended release; HydromorphContin; Oxycodone controlled release; morphine sulphate sustained release; morphine slow release
  Arms: Shortened interval extended release opioid
Drug: Extended Release Opioid Formulation, Standard intervals — Extended release opioid, individualized total daily dose, dosing interval is every 12 hours
  Other Names: Hydromorphone extended release; HydromorphContin; Oxycodone controlled release; Morphine sulphate sustained release; morphine slow release
  Arms: Standard interval extended release opioid
Drug: Placebo oral tablet — Lactose pill manufactured to mimic extended release opioid formulation
  Other Names: Placebo (for Extended release opioid)

SUMMARY:
This study is to determine the feasibility of an n-of-1, randomized, double blind, placebo controlled case series to examine effects of extended release opioids when used at intervals shorter than recommended by the manufacturer by people with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* willing and capable to give written informed consent
* diagnosis of chronic pain (> 3 months)
* current prescription for oxycodone controlled release or hydromorphone controlled release or morphine sustained release for pain
* Using extended release opioids at intervals less than 12 hours/ more than twice daily

Exclusion Criteria:

* ongoing acute pain episode
* use of immediate release opioids that contribute to more than 20% of their total daily opioid dose
* total daily morphine equivalent dose >400mg
* actively tapering their opioid dose
* use of multiple extended release opioid products
* unstable psychological diagnosis (using the Psychosocial Screening Interview Guide)
* outstanding or planned litigation related to pain
* pregnancy or lactation in women
* history of coronary artery disease
* active tapering or titration of benzodiazepines or cannabinoids
* positive urine drug screen for amphetamines, barbiturates, cocaine, methamphetamine, methadone, phencyclidine, propoxyphene or unexpected opioids or benzodiazepines
* using M-Eslon
* using long acting hydromorphone
* using Kadian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-03-08 (Actual); Study Completion 2020-03-08 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who complete both treatment periods and have evaluable Patient Global Impression and pharmacokinetic data | 8 months
  Feasibility outcome

SECONDARY OUTCOMES:
Patient Global Impression of Change | 3 weeks
  Single-item rating by subjects of their improvement with treatment on a 7-point scale that ranges from the lowest rating of 1= 'very much improved' to the highest rating of 7= 'very much worse'. Higher values are considered to be a better outcome.
Numerical Pain Rating Scale | 3 weeks
  A measure of pain intensity. Ten point scale with a minimum of "0"= no pain to a maximum of "10" = worst pain imaginable. Higher scores represent a worse outcome.
Brief Pain Inventory (Short Form) | 3 weeks
  An inventory of questions about pain, including a pain diagram, pain intensity rating subscales and pain interference rating subscales. The four pain intensity rating subscales are "pain at worst", "pain at least", "pain on average" and "pain right now". These are 10-point scales with a minimum of "0" =no pain, and a maximum of "10"= pain as bad as you can imagine", where higher scores are worse. Pain intensity subscales can be combined as an average on the same scale of 0-10. The eight pain interference subscales measuring interference on general activity, mood, walking ability, work, relations with other people, sleep, enjoyment of life, are 10-point subscales which range a minimum of "0" = pain does not interfere, to a maximum of "10"=pain completely interferes with the item. Higher scores are worse outcomes. Pain interference subscales may be combined as an total score out of 80, or divided by eight to get an average of pain interference on the scale of 0-10.
Subjective Opioid Withdrawal Scale | 3 weeks
  A self-administered scale for grading 16 opioid withdrawal symptoms on a scale of '0' meaning 'not at all' to '4' meaning 'extremely'. Higher numbers are worse outcomes.
Addiction Research Centre Inventory (ARCI) - short form | 8 hours
  The short version of the ARCI is a well-validated, standardized, self-report questionnaire of 49 "true-false" items and is used to differentiate subjective effects of drugs. True = 1, False = 0, responses to selected items are added for scores on different scales. Three of the scales are pertinent to opioid abuse liability: MBG (morphine-benzedrine group), a measure of euphoria, minimum = 0, and a maximum = 16); PCAG (pentobarbital-chlorpromazine-alcohol group) a measure of sedation, minimum =0, maximum=15; LSD (lysergic acid diethylamide scale) a measure of dysphoric and psychotomimetic changes, minimum=0, maximum =14. Higher scores are worse outcomes.
Profile of Mood States | 8 hours
  A widely used, self-reported questionnaire for assessing drug-induced changes in mood. It has 72 adjectives and phrases describing feelings people have, and ask for the user to describe "how you are feeling right now" on a 5 point scale of descriptives: with a minimum value = 0 "Not at all", to a maximum value of 4= "extremely". Total mood disturbance is calculated by adding the results of the 6 subscales, and then subtracting the vigor -activity subscale (range 0-200). Subscales (six) are calculating by adding specific items: tension-anxiety (9 items, range 0-36), depression (15 items, range 0-60), anger-hostility (12 items, range 0-48), vigor-activity (8 items, range 0-32), fatigue (7 items, range 0-28), confusion-bewilderment (7 items, range 0-28).
Visual analogue scale - liking/high | 8 hours
  Visual analog scales are 100mm lines, anchored at the ends by opposing adjectives (e.g. like-dislike). "Like" is at the minimum, 0mm mark, "dislike" is at the maximum, 100mm mark. Subjects are instructed to rate how they feel along a continuum by making a mark along the line. The measurement of drug liking is considered to be one of the most sensitive and reliable assessments of the likelihood of abuse of a drug. "Liking" and "High" at the 100mm marks would be considered worse outcomes in terms of likelihood of abuse of a substance.
Serum opioid concentrations | 6 hours
  Serum opioid concentrations at 0,30 mins, 1,2,3,4,5,6 hours post-dose
Peak plasma concentration (Cmax) | 6 hours
  The maximum concentration achieved post dose
Time to peak plasma concentration (Tmax) | 6 hours
  Time that peak plasma concentration occurs post-dose
Area under the plasma concentration versus time curve (AUC) | 24 hours
  Calculated area under the plasma concentration versus time curve, which describes exposure to the drug.
Abuse liability quotient (AQ) | 6 hours
  The peak plasma concentration (Cmax) divided by the time to peak plasma concentration, which describes a calculation of the average rate of increase in plasma concentration over the interval between treatment administration and the time of peak plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Furlan, MD, PhD, Principal Investigator — Principal Investigator
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No